CLINICAL TRIAL: NCT03144596
Title: The Effects of Systemic Alfuzosin and Tamsulosin Hydrochloride on Choroidal Thickness and Pupil Diameter Sizes in Cases With Benign Prostatic Hyperplasia
Brief Title: The Effects of α-adrenergic Receptor Antagonists on Choroid and Pupil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocatepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-KAEK-2 2015/342
Record Dates: First submitted 2017-05-02; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Benign Prostatic Hyperplasia; Pupil Anomaly; Choroid Disease
MeSH Terms: conditions — Prostatic Hyperplasia; Pupil Disorders; Choroid Diseases | interventions — alfuzosin; Tamsulosin

STUDY DESIGN:
Intervention Model Description: prospective, randomized, parallel-group clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alfuzosin Hydrochloride (Experimental): Alfuzosin hydrochloride 10 mg tablet by mouth, every 24 hours for 3 months
  Interventions: Drug: Alfuzosin Hydrochloride 10 MG
- Tamsulosin Hydrochloride (Active Comparator): Tamsulosin hydrochloride 0.4 mg tablet by mouth, every 24 hours for 3 months
  Interventions: Drug: Tamsulosin Hydrochloride 0.4 MG

INTERVENTIONS:
Drug: Alfuzosin Hydrochloride 10 MG — Alfuzosin hydrochloride Tablet
  Other Names: Xatral
  Arms: Alfuzosin Hydrochloride
Drug: Tamsulosin Hydrochloride 0.4 MG — Tamsulosin Hydrochloride Tablet
  Other Names: Flomax
  Arms: Tamsulosin Hydrochloride

SUMMARY:
It was aimed to evaluate and investigate the effects of tamsulosin hydrochloride, has preferential selectivity for the α1A receptor in the prostat versus the α1B receptor in the blood vessels, and alfuzosin hydrochloride on choroidal thickness (CT), pupil diameter sizes evaluated by using enhanced depth imaging spectral-domain optical coherence tomography (EDI-OCT) and scheimpflug/placido photography-based topoghraphy system in this study.

63 men patients with newly diagnosis of benign prostatic hyperplasia were randomly assigned to either alfuzosin hydrochloride or to tamsulosin hydrochloride groups in this prospective, randomized, parallel-group clinical trial. Enhanced depth imaging spectral-domain optical coherence tomography, pupillography were obtained at baseline, 1st and 3rd month, and choroidal thicknesses and pupil diameter sizes were compared between the 2 groups.

DETAILED DESCRIPTION:
The local authorized clinical trials ethics committee approved the study and this study was performed following the principles of the Declaration of Helsinki. Detailed information was given to patients about clinical applications and tests, and signed informed consent forms were also obtained from all patients. 32 right eyes of 32 men with diagnosis of BPH initiated on AH (Xatral®) (10 mg/day) and 31 right eyes of 31 men with diagnosis of BPH initiated on TH (Flomax®) (0.4 mg/day) were included in this self-controlled prospective clinical trial. Urologists in the urology clinic made diagnosis of BPH, and 63 men diagnosis of BPH were directed towards eye clinic. AH or TH treatments were randomly recommended for previously untreated patients with newly diagnosis of BPH by urologists. After providing information to patients about the disease and treatment, patients predicted to show adherence to treatment, were enrolled in the study.

Ophthalmological examinations were performed in all cases. Choroidal thicknesses (CTs) were measured under the fovea, 3 mm nasal to the fovea and 3 mm temporal to the fovea, and they were recorded as submacular (SCT), nasal (NCT) and temporal (TCT) choroidal thicknesses. CTs were measured and recorded by using EDI-OCT imaging (Cirrus HD 4000, Carl Zeis Meditec, CA, USA). Mesopic, scotopic and photopic pupil diameter sizes were measured and recorded by using Scheimpflug/Placido photography-based topography system in the pupillometer mode (Sirius, Italy). CTs, scotopic, mesopic and photopic pupil diameter sizes were measured and recorded at baseline, 1st and 3rd months.

Data obtained from cases were encoded and they were transferred to the computer program. SPSS 20.0 software (SPSS Inc., Chicago, IL, USA) was used for statistical evaluation. Data distribution was tested using Kolmogorov-Smirnov test. Baseline values and 1st, 3rd month values were compared by using the repeated measure of ANOVA in intra-group evaluation and independent samples t-test in inter-group evaluation, and the significance level of p-value was accepted as 0,05 (P ≤ 0, 05). Progressions were evaluated by using repeated measures analyses of variance-ANOVA (with the Bonferroni correction) and the correlation between parameters were evaluated by using bivariate (Pearson's) correlation analysis. Positive values and negative values were considered to be correlated in the same direction and opposite direction, respectively in correlation analysis. Correlation coefficient values r ≥ |± 0.3| were accepted as correlation; and the significance level of P value that was below 0,05 was evaluated as the significant correlation.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity (BCVA) ≥ 0.8
* Diagnosis of BPH and initiation of alfuzosin hydrochloride or tamsulosin hydrochloride treatments
* 45 years of age or older man

Exclusion Criteria:

* Occluded angle by gonioscopy (grade 0, narrow angle, grade I, grade II)
* Corneal scarring or cataract that prevents appearance of the fundus
* Formation of macular or peripheral retinal pathologies or choroidopathy
* Optic nerve pathologies such as optic neuropathy
* Spherical refractive error ≥ ±6.00 D or cylinder refractive error ≥ ±3.00 D
* Systemic diseases that may affect choroidal blood flow

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 63 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2016-11-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline choroidal thicknesses at 3 months | 1 month and 2 months
  Choroidal thicknesses (CTs) measurement under the fovea, 3 mm nasal to the fovea and 3 mm temporal to the fovea at baseline, 1st and 3rd month, and recording as submacular (SCT), nasal (NCT) and temporal (TCT) choroidal thicknesses.
Change from baseline pupil diameter sizes at 3 months | 1 month and 2 months
  Mesopic, scotopic and photopic pupil diameter sizes measurement at baseline, 1st and 3rd months

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Dogan, Asst. Prof., Study Director — Afyon Kocatepe University Eye Clinics

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berry SJ, Coffey DS, Walsh PC, Ewing LL. The development of human benign prostatic hyperplasia with age. J Urol. 1984 Sep;132(3):474-9. doi: 10.1016/s0022-5347(17)49698-4. PMID 6206240
- [Background] Yuan J, Liu Y, Yang Z, Qin X, Yang K, Mao C. The efficacy and safety of alpha-1 blockers for benign prostatic hyperplasia: an overview of 15 systematic reviews. Curr Med Res Opin. 2013 Mar;29(3):279-87. doi: 10.1185/03007995.2013.766594. Epub 2013 Jan 29. PMID 23323875
- [Background] McVary KT, Roehrborn CG, Avins AL, Barry MJ, Bruskewitz RC, Donnell RF, Foster HE Jr, Gonzalez CM, Kaplan SA, Penson DF, Ulchaker JC, Wei JT. Update on AUA guideline on the management of benign prostatic hyperplasia. J Urol. 2011 May;185(5):1793-803. doi: 10.1016/j.juro.2011.01.074. Epub 2011 Mar 21. PMID 21420124
- [Background] Filson CP, Hollingsworth JM, Clemens JQ, Wei JT. The efficacy and safety of combined therapy with alpha-blockers and anticholinergics for men with benign prostatic hyperplasia: a meta-analysis. J Urol. 2013 Dec;190(6):2153-60. doi: 10.1016/j.juro.2013.05.058. Epub 2013 May 30. PMID 23727412
- [Background] Osman NI, Chapple CR, Cruz F, Desgrandchamps F, Llorente C, Montorsi F. Silodosin : a new subtype selective alpha-1 antagonist for the treatment of lower urinary tract symptoms in patients with benign prostatic hyperplasia. Expert Opin Pharmacother. 2012 Oct;13(14):2085-96. doi: 10.1517/14656566.2012.714368. Epub 2012 Aug 28. PMID 22924980
- [Background] Oelke M, Gericke A, Michel MC. Cardiovascular and ocular safety of alpha1-adrenoceptor antagonists in the treatment of male lower urinary tract symptoms. Expert Opin Drug Saf. 2014 Sep;13(9):1187-97. doi: 10.1517/14740338.2014.936376. Epub 2014 Jul 29. PMID 25073735
- [Background] Hollingsworth JM, Wilt TJ. Lower urinary tract symptoms in men. BMJ. 2014 Aug 14;349:g4474. doi: 10.1136/bmj.g4474. PMID 25125424
- [Background] Schwinn DA, Michelotti GA. alpha1-adrenergic receptors in the lower urinary tract and vascular bed: potential role for the alpha1d subtype in filling symptoms and effects of ageing on vascular expression. BJU Int. 2000 Apr;85 Suppl 2:6-11. doi: 10.1046/j.1464-410x.2000.00061.x. No abstract available. PMID 10781179
- [Background] Hatano A, Takahashi H, Tamaki M, Komeyama T, Koizumi T, Takeda M. Pharmacological evidence of distinct alpha 1-adrenoceptor subtypes mediating the contraction of human prostatic urethra and peripheral artery. Br J Pharmacol. 1994 Nov;113(3):723-8. doi: 10.1111/j.1476-5381.1994.tb17053.x. PMID 7858860
- [Background] de Mey C. alpha(1)-blockers for BPH: are there differences? Eur Urol. 1999;36 Suppl 3:52-63. doi: 10.1159/000052349. PMID 10559631
- [Background] Dunn CJ, Matheson A, Faulds DM. Tamsulosin: a review of its pharmacology and therapeutic efficacy in the management of lower urinary tract symptoms. Drugs Aging. 2002;19(2):135-61. doi: 10.2165/00002512-200219020-00004. PMID 11950378
- [Background] Bird ST, Delaney JA, Brophy JM, Etminan M, Skeldon SC, Hartzema AG. Tamsulosin treatment for benign prostatic hyperplasia and risk of severe hypotension in men aged 40-85 years in the United States: risk window analyses using between and within patient methodology. BMJ. 2013 Nov 5;347:f6320. doi: 10.1136/bmj.f6320. PMID 24192967
- [Background] Chrischilles E, Rubenstein L, Chao J, Kreder KJ, Gilden D, Shah H. Initiation of nonselective alpha1-antagonist therapy and occurrence of hypotension-related adverse events among men with benign prostatic hyperplasia: a retrospective cohort study. Clin Ther. 2001 May;23(5):727-43. doi: 10.1016/s0149-2918(01)80022-9. PMID 11394731
- [Background] Chang DF, Campbell JR. Intraoperative floppy iris syndrome associated with tamsulosin. J Cataract Refract Surg. 2005 Apr;31(4):664-73. doi: 10.1016/j.jcrs.2005.02.027. PMID 15899440
- [Background] Abdel-Aziz S, Mamalis N. Intraoperative floppy iris syndrome. Curr Opin Ophthalmol. 2009 Jan;20(1):37-41. doi: 10.1097/ICU.0b013e32831bc0ad. PMID 19077827
- [Background] Mamalis N. Intraoperative floppy-iris syndrome associated with systemic alpha blockers. J Cataract Refract Surg. 2008 Jul;34(7):1051-2. doi: 10.1016/j.jcrs.2008.05.017. No abstract available. PMID 18571055
- [Background] Chang DF, Braga-Mele R, Mamalis N, Masket S, Miller KM, Nichamin LD, Packard RB, Packer M; ASCRS Cataract Clinical Committee. ASCRS White Paper: clinical review of intraoperative floppy-iris syndrome. J Cataract Refract Surg. 2008 Dec;34(12):2153-62. doi: 10.1016/j.jcrs.2008.08.031. PMID 19027575
- [Background] Nickla DL, Wallman J. The multifunctional choroid. Prog Retin Eye Res. 2010 Mar;29(2):144-68. doi: 10.1016/j.preteyeres.2009.12.002. Epub 2009 Dec 29. PMID 20044062
- [Background] Konno F, Takayanagi I. Characterization of postsynaptic alpha 1-adrenoceptors in the rabbit iris dilator smooth muscle. Naunyn Schmiedebergs Arch Pharmacol. 1986 Jul;333(3):271-6. doi: 10.1007/BF00512940. PMID 2876390
- [Background] Shapiro BL, Petrovic V, Lee SE, Flach A, McCaffery S, O'Brien JM. Choroidal detachment following the use of tamsulosin (Flomax). Am J Ophthalmol. 2007 Feb;143(2):351-3. doi: 10.1016/j.ajo.2006.09.032. Epub 2006 Oct 23. PMID 17258532
- [Background] Kerimoglu H, Zengin N, Ozturk B, Gunduz K. Unilateral chemosis, acute onset myopia and choroidal detachment following the use of tamsulosin. Acta Ophthalmol. 2010 Mar;88(2):e20-1. doi: 10.1111/j.1755-3768.2008.01503.x. Epub 2009 Mar 19. No abstract available. PMID 19302075
- [Background] Nieminen T, Ylitalo R, Koobi T, Ylitalo P, Kahonen M. The vasodilatory effect of alfuzosin and tamsulosin in passive orthostasis: a randomised, double-blind, placebo-controlled study. Eur Urol. 2005 Mar;47(3):340-5. doi: 10.1016/j.eururo.2004.11.002. Epub 2004 Dec 29. PMID 15716198
- [Background] Gu N, Kim J, Lim KS, Shin KH, Kim TE, Lee B, Shin SG, Jang IJ, Yu KS. Assessment of the effect of mirodenafil on the hemodynamics of healthy male Korean volunteers administered tamsulosin: a randomized, double-blind, placebo-controlled, 2-period crossover study. Clin Ther. 2012 Sep;34(9):1929-39. doi: 10.1016/j.clinthera.2012.08.002. Epub 2012 Aug 24. PMID 22921287
- [Background] Kiel JW, Lovell MO. Adrenergic modulation of choroidal blood flow in the rabbit. Invest Ophthalmol Vis Sci. 1996 Mar;37(4):673-9. PMID 8595968
- [Background] Tanabe H, Ito Y, Iguchi Y, Ozawa S, Ishikawa K, Terasaki H. Correlation between cross-sectional shape of choroidal veins and choroidal thickness. Jpn J Ophthalmol. 2011 Nov;55(6):614-9. doi: 10.1007/s10384-011-0079-2. Epub 2011 Aug 27. PMID 21874308
- [Background] Vance SK, Imamura Y, Freund KB. The effects of sildenafil citrate on choroidal thickness as determined by enhanced depth imaging optical coherence tomography. Retina. 2011 Feb;31(2):332-5. doi: 10.1097/IAE.0b013e3181eef0ae. PMID 20975620